CLINICAL TRIAL: NCT06206174
Title: A Single-arm, Open-label, Dose Escalation and Expansion Phase I/II Study Evaluating Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of TGRX-814 Monotherapy and Combination Therapy in Patients With Hematological Malignancies
Brief Title: TGRX-814 Chinese Phase I/II in Patients With Hematological Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen TargetRx, Inc. (Industry)
Collaborators: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGRX-814-1001
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Hematologic Malignancy; Non Hodgkin Lymphoma; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia, Adult; Myelodysplastic Syndromes
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma, Non-Hodgkin; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TGRX-814 (Experimental): TGRX-814 monotherapy for Dose escalation study; oral, once daily administration.
  Interventions: Drug: TGRX-814

INTERVENTIONS:
Drug: TGRX-814 — Participants are given TGRX-814 tablets for oral, once daily administration at one of the dose levels as pre-determined for the dose escalation sequence.
  Other Names: TGRX-814 monotherapy

SUMMARY:
The purpose of this single- arm, open-label, dose escalation and dose expansion phase I/II study is to evaluate the safety, tolerability, pharmacokinetic and preliminary efficacy of TGRX-814 in patients with hematological malignancies including non-Hodgkin lymphoma, acute myeloid leukemia, aute lymphoblastic leukemia and myelodysplastic syndromes.

DETAILED DESCRIPTION:
This is the first-in-human trial with TGRX-814 which aims to evaluate the safety, pharmacokinetic and preliminary efficacy profiles with hematological malignancies. The primary purpose of this study is to evaluate the safety profile of TGRX-814 in patients with non-Hodgkin lymphoma and to determine of the maximal tolerated dose (MTD) and recommended phase II dose (RP2D). Other purposes of the study include evaluating safety and preliminary efficacy of TGRX-814 monotherapy and combination therapy in patients with other types of hematological malignancies, including acute myeloid leukemia, aute lymphoblastic leukemia and myelodysplastic syndromes, as well as evaluating the pharmacokinetic profile of TGRX-814. The study is a phase I/II study, consisting a monotherapy dose escalation study, monotherapy dose expansion study and combination therapy study.

ELIGIBILITY:
Inclusion Criteria:

1. male or female ≥ 18 years of age
2. fully understand the requirements of the study and voluntarily sign a written informed consent form
3. diagnosis of NHL, ALL, AML or MDS
4. Eastern Cooperative Oncology Group (ECOG) physical status score ≤ 2
5. adequate bone marrow function
6. patients at high risk for Tumor Lysis Syndrome (TLS) determined by investigator and sponsor for agreement to enroll
7. adequate disease indicator
8. adequate coagulation, hepatic and renal function
9. female subjects of childbearing potential and male subjects whose partners are women of childbearing potential must agree to use a medically approved highly effective contraceptive from the time of signing the Informed Consent Form until at least 3 months after the last dose of study drug; women of childbearing potential must have a negative blood or urine pregnancy test within 7 days prior to the first dose of study drug
10. Expected survival time ≥ 12 weeks

Exclusion Criteria:

1. received BCL-2 inhibitor therapy prior to the first dose of study drug, unless discontinued due to intolerance
2. subjects with NHL have been diagnosed with Burkitt's lymphoma, lymphoblastoid lymphoma/leukemia, or post-transplant lymphoproliferative disease (PTLD)
3. AML subjects with a diagnosis of acute promyelocytic leukemia or Ph chromosome positive or persistent extramedullary leukemia
4. tumor infiltration of the central nervous system
5. received allogeneic hematopoietic stem cell transplantation; or received autologous hematopoietic stem cell transplantation within 3 months
6. received vaccination within 4 weeks prior to first dose or scheduled to be vaccinated during the study
7. HBsAg-positive or HBcAb-positive; HCV antibody-positive; HIV antibody-positive
8. monoclonal antibody antitumor therapy within 4 weeks prior to the first dose; participation in a clinical trial of another interventional drug within 4 weeks prior to the first dose; participation in CAR-T therapy within 12 weeks prior to the first dose; 9. 14 weeks prior to the first dose
9. received anticancer therapy/investigational therapy within 14 days prior to the first dose, or has not recovered from clinically significant toxicity below grade 2 on prior therapy
10. received steroidal anticancer therapy, CYP3A inhibitors, or CYP3A inducers within 7 days prior to the first dose of study drug
11. consumption of grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges), or popcorn within 3 days prior to the first dose of the drug
12. poorly controlled hypertension; left ventricular ejection fraction ≤ 50% as assessed by cardiac ultrasound; prolonged QT interval; Grade III atrioventricular block or other arrhythmia requiring medical intervention; New York Heart Association (NYHA) Class III or IV congestive heart failure; had myocardial infarction or experienced bypass surgery within 6 months prior to dosing; had arterial or venous thrombotic events within 6 months prior to the first dose of study drug; have other cardiovascular diseases that investigator deemed unfit for enrollment
13. having a history of renal, neurological, psychiatric, pulmonary, endocrine, metabolic, immunologic, cardiovascular, or hepatic disease that, in the opinion of the Investigator, would adversely affect the subject's participation in this study
14. having a history of active malignancy other than NHL, AML, or MDS within 3 years prior to participation in this clinical study
15. having a condition of malabsorption syndrome or multiple factors that interfere with the oral administration and absorption of medication
16. other uncontrolled conditions of clinical significance
17. other factors that, in the opinion of the Investigator, may affect the results of the study and interfere with the patient's participation in the study, including previous or existing medical conditions, abnormalities in treatment or laboratory tests, unwillingness of the subject to comply with the procedures, restrictions and requirements of the study, and other conditions that make enrollment in the study unsuitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Maximal tolerated dose (MTD) | At end of dose escalation when the probability of DLT of a dose level is greater than 0.359
  To determine the MTD of TGRX-814 in non-Hodgkin lymphoma (NHL) patients
Recommended phase II dose (RP2D) | At completion of the dose escalation study, an average of 1 year
  To determine the RP2D of TGRX-814 in NHL patients for Phase II

SECONDARY OUTCOMES:
Dose-limiting toxicities (DLTs) | DLT is collected during Cycle 1 (each cycle is 28 days)
  to record and analyze DLTs in all patients with hematological malignancies
Adverse Events (AEs)/Serious Adverse Events (SAEs) | AE and SAE are collected throughout and until completion of the study, an average of 1 year.
  to record and analyze AEs/SAEs in all patients with hematological malignancies
Complete Response (CR) rate | at screening period, at the end of week 8, 16, 24, 36, 48, subsequent every 24 weeks and the last visit of treatment period, at the end-of-treatment follow-up visit and safety follow-up visit
  to record and analyze the CR rate in patients with NHL, ALL, AML, and MDS
Complete response with incomplete count recovery (CRi) rate | at screening period, at the end of week 8, 16, 24, 36, 48, subsequent every 24 weeks and the last visit of treatment period, at the end-of-treatment follow-up visit and safety follow-up visit
  to record and analyze the CRi rate in patients with NHL, ALL, and AML
Partial response (PR) rate | at screening period, at the end of week 8, 16, 24, 36, 48, subsequent every 24 weeks and the last visit of treatment period, at the end-of-treatment follow-up visit and safety follow-up visit
  to record and analyze the PR rate in patients with NHL, AML, and MDS
Partial response with lymphocytosis (PRL) rate | at screening period, at the end of week 8, 16, 24, 36, 48, subsequent every 24 weeks and the last visit of treatment period, at the end-of-treatment follow-up visit and safety follow-up visit
  to record and analyze the PRL rate in patients with NHL
Stable disease (SD) rate | at screening period, at the end of week 8, 16, 24, 36, 48, subsequent every 24 weeks and the last visit of treatment period, at the end-of-treatment follow-up visit and safety follow-up visit
  to record and analyze the SD rate in patients with NHL
Objective response rate (ORR) | at screening period, at the end of week 8, 16, 24, 36, 48, subsequent every 24 weeks and the last visit of treatment period, at the end-of-treatment follow-up visit and safety follow-up visit
  to record and analyze the ORR in patients with NHL
Duration of complete response (DCR) | at screening period, at the end of week 8, 16, 24, 36, 48, subsequent every 24 weeks and the last visit of treatment period, at the end-of-treatment follow-up visit and safety follow-up visit
  to record and analyze the DCR in patients with NHL and AML
Duration of response (DOR) | at screening period, at the end of week 8, 16, 24, 36, 48, subsequent every 24 weeks and the last visit of treatment period, at the end-of-treatment follow-up visit and safety follow-up visit
  to record and analyze the DOR in patients with NHL, ALL, AML and MDS
Overall Survival (OS) rate | at screening period, at the end of week 8, 16, 24, 36, 48, subsequent every 24 weeks and the last visit of treatment period, at the end-of-treatment follow-up visit and safety follow-up visit
  to record and analyze the OS rate in patients with NHL, ALL, AML and MDS
Morphologic leukemia-free state (MLFS) rate | at screening period, at the end of week 8, 16, 24, 36, 48, subsequent every 24 weeks and the last visit of treatment period, at the end-of-treatment follow-up visit and safety follow-up visit
  to record and analyze the MLFS rate in patients with ALL and AML
Complete response with partial hematologic recovery (CRh) | at screening period, at the end of week 8, 16, 24, 36, 48, subsequent every 24 weeks and the last visit of treatment period, at the end-of-treatment follow-up visit and safety follow-up visit
  to record and analyze the CRh rate in patients with ALL
Molecular complete response (mCR) rate | at screening period, at the end of week 8, 16, 24, 36, 48, subsequent every 24 weeks and the last visit of treatment period, at the end-of-treatment follow-up visit and safety follow-up visit
  to record and analyze the mCR rate in patients with MDS
Progress-Free survival (PFS) rate | at screening period, at the end of week 8, 16, 24, 36, 48, subsequent every 24 weeks and the last visit of treatment period, at the end-of-treatment follow-up visit and safety follow-up visit
  to record and analyze the PFS rate in patients withAML
Minimum concentration at steady state (Css-min) | at screening period, and at day 1, 15 and 22 of Cycle 1, day 1 of Cycle 3, day 1 of Cycle 5, and day 1 of Cycle 7 of the treatment period (each Cycle is 28 days)
  to measure/calculate the Pharmacokinetic (PK) parameter of Css-min in all patients with hematological malignancy
Maximum concentration at steady state (Css-max) | at screening period, and at day 1, 15 and 22 of Cycle 1, day 1 of Cycle 3, day 1 of Cycle 5, and day 1 of Cycle 7 of the treatment period (each Cycle is 28 days)
  to measure/calculate the PK parameter of Css-max in all patients with hematological malignancy
Average concentration at steady state (Css-ave) | at screening period, and at day 1, 15 and 22 of Cycle 1, day 1 of Cycle 3, day 1 of Cycle 5, and day 1 of Cycle 7 of the treatment period (each Cycle is 28 days)
  to measure/calculate the PK parameter of Css-ave in all patients with hematological malignancy
Time of Maximum concentration at steady state (Tmax,ss) | at screening period, and at day 1, 15 and 22 of Cycle 1, day 1 of Cycle 3, day 1 of Cycle 5, and day 1 of Cycle 7 of the treatment period (each Cycle is 28 days)
  to measure/calculate the PK parameter of Tmax,ss in all patients with hematological malignancy
Area-under-curve in treatment interval at steady state (AUCtau-ss) | at screening period, and at day 1, 15 and 22 of Cycle 1, day 1 of Cycle 3, day 1 of Cycle 5, and day 1 of Cycle 7 of the treatment period (each Cycle is 28 days)
  to measure/calculate the PK parameter of AUCtau-ss in all patients with hematological malignancy
Volume of distribution at steady state (Vss) | at screening period, and at day 1, 15 and 22 of Cycle 1, day 1 of Cycle 3, day 1 of Cycle 5, and day 1 of Cycle 7 of the treatment period (each Cycle is 28 days)
  to measure/calculate the PK parameter of Vss in all patients with hematological malignancy
Accumulation ratio (AR) | at screening period, and at day 1, 15 and 22 of Cycle 1, day 1 of Cycle 3, day 1 of Cycle 5, and day 1 of Cycle 7 of the treatment period (each Cycle is 28 days)
  to measure/calculate the PK parameter of AR in all patients with hematological malignancy
Degree of fluctuation (DF) | at screening period, and at day 1, 15 and 22 of Cycle 1, day 1 of Cycle 3, day 1 of Cycle 5, and day 1 of Cycle 7 of the treatment period (each Cycle is 28 days)
  to measure/calculate the PK parameter of DF in all patients with hematological malignancy

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China; Bo Jiang, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China